CLINICAL TRIAL: NCT01003574
Title: Evaluation of Cardiovascular Health Outcomes Among Survivors
Acronym: ECHOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ECHOS; R01NR011322 (NIH)
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Cardiovascular Risk; Cancer
Keywords: cardiovascular health outcomes in cancer survivors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Other): Control arm will receive standard care for risk of cardiac sequelae - a mailed, tailored (neither generic nor targeted) print summary of individualized information about the survivor's treatment, late effects risks, and recommended follow-up and lifestyle modifications.
  Interventions: Behavioral: lifestyle modification and telephone counseling
- Test Arm (Other): Test arm will receive standard care plus motivational, autonomy-supportive APN counseling (2 phone sessions) that targets two categories of behavioral constructs likely to influence screening.
  Interventions: Behavioral: lifestyle modification and telephone counseling

INTERVENTIONS:
Behavioral: lifestyle modification and telephone counseling — A mailed individualized cancer treatment summary with recommendations for CV follow-up and lifestyle modification (standard care).
  Other Names: Cardiovascular Health Outcomes
  Arms: Control Arm
Behavioral: lifestyle modification and telephone counseling — Standard care plus motivational, autonomy-supportive APN counseling (2 phone sessions) that targets two categories of behavioral constructs likely to influence screening.
  Other Names: Cardiovascular Health Outcomes
  Arms: Test Arm

SUMMARY:
This study will test a 2-tiered tailored intervention and evaluation of cardiovascular health outcomes among survivors designed to inform childhood cancer survivors about their individual cardiac risk and follow-up recommendations and to provide motivational support for cardiovascular (CV) screening. This study will test if the addition of telephone motivational interviewing, tailored to behavioral constructs, is superior to the current standard of care in increasing survivors' CV screening.

DETAILED DESCRIPTION:
* This study will test the hypothesis that at 1 year post-intervention, a significantly greater proportion of the advanced-practice nurse (APN) phone counseling group will have undergone cardiovascular screening, as compared to the standard care group. Cardiovascular (CV) screening will be defined, based on established CV screening recommendations, as completion of an imaging evaluation of left ventricular systolic function (i.e., echocardiogram, multiple uptake gated acquisition scan, or cardiac magnetic resonance imaging).
* This study will measure changes induced by the intervention in survivors' knowledge, motivation, fear, beliefs, affect, readiness for medical follow-up, and self-efficacy and these changes' potential mediating effects on CV screening.

  * This study will provide a cost analysis of the ECHOS intervention in terms of the cost of left ventricular systolic function imaging per additional survivor screened, an estimate of the cost of standard care per survivor screened, and the cost of screening and follow-up per survivor screened.

ELIGIBILITY:
Inclusion Criteria:

1. Childhood Cancer Survivor Study (CCSS) cohort participants
2. Age 25 years or older
3. No CV screening in previous 5 years
4. Received anthracycline chemotherapy and/or irradiation of the chest
5. Previous history of successful independent (non-surrogate) response to CCSS surveys (reading level for non-medical items is 4th-6th grade Flesch-Kincaid level).

Exclusion Criteria:

1. Being followed at an institution actively recruiting adults to a long-term follow-up program (ascertained in CCSS follow-up database)
2. Inability or unwillingness of research participant to give written informed consent.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2010-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
This study will test the hypothesis that at 1 year post-intervention, a significantly greater proportion of the APN phone counseling group will have undergone cardiovascular screening, as compared to the standard care group | 2.5 years

SECONDARY OUTCOMES:
Change in knowledge | Baseline and 2.5 years post intervention
Change in motivation | Baseline and 2.5 years post intervention
Change in fear | Baseline and 2.5 years post intervention
Change in beliefs | Baseline and 2.5 years post intervention
Change in affect | Baseline and 2.5 years post intervention
Change in readiness for medical follow-up | Baseline and 2.5 years post intervention
Change in self-efficacy | Baseline and 2.5 years post intervention
Estimated average cost of intervention per participant | 2.5 years
Estimated average cost of standard care per participant in the Control Arm | 2.5 years
Estimated average cost of cardiovascular screening per participant in the Test Arm | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Hudson, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Hudson MM, Leisenring W, Stratton KK, Tinner N, Steen BD, Ogg S, Barnes L, Oeffinger KC, Robison LL, Cox CL. Increasing cardiomyopathy screening in at-risk adult survivors of pediatric malignancies: a randomized controlled trial. J Clin Oncol. 2014 Dec 10;32(35):3974-81. doi: 10.1200/JCO.2014.57.3493. Epub 2014 Nov 3. PMID 25366684
- See also: St. Jude Children's Research Hospital — http://www.stjude.org